CLINICAL TRIAL: NCT06967350
Title: Research on the Construction and Application of a New Model of Outpatient Nurse-Patient Communication Based on CARE Combined With AIDET and Service Recovery Theory
Brief Title: Research on the Application of CARE Combined With AIDET Nurse-Patient Communication Model in Implementing Service Remediation in Outpatient Clinics
Acronym: CARE AIDET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bao Yan (Other)
Responsible Party: Sponsor-Investigator, Bao Yan, Deputy Director, The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Organization: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KY-2024-023
Record Dates: First submitted 2025-05-12; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Communication; Service Recovery
Keywords: CARE; AIDET
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group 1(CARE training) (Other): This study adopted a parallel control design and set up the CARE group as the control group 1. The nurses in this group received training on the CARE communication model: including theoretical lectures, case discussions, pre-operation practical assessment, and clinical pre-operation practical supervision.
  Interventions: Other: CARE communication mode
- control group 2(AIDET training) (Other): This study adopted a parallel control design and set up the AIDET group as the control group 2. The nurses in this group received AIDET communication mode training: including theoretical lectures, case discussions, pre-operation practical assessment, and clinical pre-operation practical supervision.
  Interventions: Other: AIDET communication mode
- Experimental Group (CARE &AIDET) (Experimental): This study adopted a parallel control design and set up the CARE&AIDET group as the experimental group. The nurses in this group received training on the CARE combined with AIDET communication model: including theoretical lectures, case discussions, pre-operation practical assessment, and clinical pre-operation practical supervision.
  Interventions: Other: CARE & AIDET communication mode

INTERVENTIONS:
Other: CARE & AIDET communication mode — The new communication mode, which incorporates fundamental communication principles (AIDET) and service recovery strategies (CARE)
  Arms: Experimental Group (CARE &AIDET)
Other: CARE communication mode — CARE (C: connect, A: apologize, R: repair, E: exceed) is a standard service recovery communication mode in medical services.
  Arms: control group 1(CARE training)
Other: AIDET communication mode — AIDET is a nurse-patient communication mode that contains essential communication principles. Each letter represents a step for communication: Acknowledge, Introduce, Duration, Explanation, and Thank. It describes in detail the application and characteristics of the primary language in communication, logical and procedural.
  Arms: control group 2(AIDET training)

SUMMARY:
CARE (C: connect, A: apologize, R: repair, E: exceed) is a standard service recovery communication mode in medical services. However, clinical nurses found it hard to follow because it lacked essential communication guidance. The AIDET mode (A: acknowledge, I: introduce, D: duration, E: Explanation, T: thank)， which offers such guidance, might be combined with CARE to form a new mode. This study aims to verify the effect of integrating CARE and AIDET on outpatient nurses' service recovery.

DETAILED DESCRIPTION:
This plan is a prospective study conducted by a certain center, aiming to explore the effect of adopting the combined communication mode of CARE and AIDET on improving the clinical communication ability of nurses when providing service remediation in outpatient care. This study strictly follows a unified research plan.

Researchers are not allowed to interfere with the clinical work of nurses. The training of communication mode education and training is arranged by the research training group. The enrolled nurses are randomly divided into three groups, and they respectively receive training in the CARE communication mode, the AIDET communication mode, and the CARE&AIDET communication mode. During the training period, nurses are allowed to learn the communication mode, including theoretical lectures, case discussions, pre-operation practical assessment, and supervision of clinical pre-operation practical operations to identify problems and raise questions. However, they are not allowed to use other communication modes and communication skills that may affect the research results to ensure the validity of the research results.

Please note that the above translation is for reference only. Specific details may vary depending on the actual situation. The observation period starts from the time the nurses are enrolled and lasts until one month after the training ends. During the entire research period, researchers closely monitor the clinical communication ability of the nurses.

This study adopts a randomized controlled trial. The focus is on evaluating the effect of the combined communication mode in the target nurse group. Data on nursing staff working in outpatient care at a certain center is collected to enhance the representativeness and reliability of the research results. At the same time, to ensure the quality of the research data, a dedicated person will be responsible for data analysis and will not participate in the project research process to ensure that the data analysis and results are not affected, and any problems in the data will be discovered and corrected.

ELIGIBILITY:
Inclusion Criteria:

* (1) nurses who have worked in the clinic for more than half a year; (2) Volunteer to participate in this study and sign a written informed consent. Unable to complete the entire study process during the study period.

Exclusion Criteria:

* (1) nurses on maternal or sick leave, rotation, or training nurses; (2)nurses with poor mental state (such as depression tendency). Therefore, we excluded rotation nurses (n=1) and maternity leave nurses (n=2) and included 75 nurses in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The score of clinical communication ability of nurses | One month before and after the training
  This score is obtained through Nurses' clinical communication ability Scale: The scale of nurses' clinical communication ability is a self-evaluation tool reflecting communication ability. The scale was developed by Zeng Kai himself and is highly recommended by Chinese scholars20. The scale has been widely used to evaluate team communication, basic verbal communication, essential non-verbal communication, emotional perception, emotional support, and difficult situation communication abilities among nurses and nursing students. The scale consists of 58 items in six dimensions. Using the Likert 5-point scale, each entry is assigned a score of 1 to 5, from "very poor" to "very good" on a scale of 58 to 290. Each entry is scored positively, and the higher the score, the better the communication ability. The Cronbach α of the scale was 0.978, and the retest reliability was 0.727.

CONTACTS AND LOCATIONS:
Locations (1):
- The fourth affiliated hospital,Zhejiang University school of medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No